CLINICAL TRIAL: NCT03638219
Title: Prognostic Significance of Bioscore in Nonmetastatic Cancer
Brief Title: Prognostic Significance of Bioscore in Nonmetastatic Breast Cancer
Acronym: Observational
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Donia Hussein Abd Elhamed, Principle invistigator, Assiut University
Other Study IDs: Bioscore in breast cancer
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection about eligible patients presented to our department from 2015 to 2018. Then follow up till 2020. — Data collection, follow up and bioscore calculation at the end of study

SUMMARY:
assess the validity of applying the bioscore system to predict the disease-free survival (The percentage of people in a study or treatment group who have not experienced disease relapse in a defined period of time.) in breast cancer patients presenting to our

DETAILED DESCRIPTION:
Retrospective cohort analysis of breast cancer patient's records for patients treated with surgery as an initial intervention at our department from 2015 to 2018 will be identified. Multivariate analyses of factors, including pathological stage (PS), T stage (T), nodal stage (N), grade (G), estrogen receptor (ER) status (E) and human epidermal growth factor receptor (HER2) status will be recorded to identify associations with disease-free survival DFS. A score of 0-4 will be assigned for each factor by considering the hazard ratio magnitude.

Analysis of the correlation between pathological stage, T stage (T), nodal stage (N), grade (G), estrogen receptor (ER) status (E) and human epidermal growth factor receptor (HER2) status combined score and the disease free survival (DFS ).

ELIGIBILITY:
Inclusion Criteria:

- Female patients Newly diagnosed breast cancer patients presented to clinical oncology department, Assiut University in the period between (2015_2018).

Histologically confirmed invasive breast carcinoma (IBC) Age: ≥18 and older Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2. Complete medical records and follow up

Exclusion Criteria:

* Male patients No definitive surgery Incomplete medical records or follow-up status Unavailability of hormonal receptor status Carcinoma in situ or other rare tumors of the breast as phylloides tumors, pregnancy and lactation

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer in female patients only.
Study Population: non metastatic breast cancer patients presenting to our department during period of our study.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
the correlation between pathological stage, T stage (T), nodal stage (N), grade (G), estrogen receptor (ER) status (E) and human epidermal growth factor receptor (HER2) status combined score and the disease specific survival (DSS) | Non metastatic breast cancer patients presented at our department from 2015 to 2018.. Then follow up till 2020
  Disease free survial:The percentage of people in a study or treatment group who have not experienced disease relapse in a defined period of time. The time period usually begins after surgerical treatment and ends at the end of study period 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Derived] Mohamed RF, Abdelhameed DH, Mohamed MA. Combination of Anatomical and Biological Factors to Predict Disease-Free Survival in Breast Cancer. JCO Glob Oncol. 2023 Mar;9:e2200269. doi: 10.1200/GO.22.00269. PMID 36888928